CLINICAL TRIAL: NCT02182791
Title: An Investigation of the Potential Pharmacokinetic Interaction Between Nevirapine (VIRAMUNE® ) and Ethinyl Estradiol/Norethindrone [ORTHO-NOVUM® 1/35 (21 Pack)] in HIV-1 Infected Women
Brief Title: Investigation of the Potential Pharmacokinetic Interaction Between Nevirapine (VIRAMUNE) and Ethinyl Estradiol/Norethindrone in HIV-1 Infected Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1100.1245
Record Dates: First submitted 2014-07-03; First posted 2014-07-08 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine

ARMS (2):
- Nevirapine tablets (Experimental): once a day (q.d.) Day 2-15,
  twice a day (b.i.d.) Study day 16-30
  Interventions: Drug: Nevirapine
- EE/NET tablets (Active Comparator): Single dose on Study Day 0 and 30
  Interventions: Drug: EE/NET

INTERVENTIONS:
Drug: Nevirapine
  Arms: Nevirapine tablets
Drug: EE/NET
  Arms: EE/NET tablets

SUMMARY:
Study to determine the effects of nevirapine treatment on the pharmacokinetics of ethinyl estradiol (EE)/norethindrone (NET).

ELIGIBILITY:
Inclusion Criteria:

* Female patients between the ages of 18 and 65 years
* Plasma HIV-1 RNA <= 400 copies/mL, documenting HIV-1 infection, within 28 days prior to Study Day 0
* Lymphocytes Expressing CD4+ Surface Marker (CD4+ cell count) >= 100 cells/mm³ within 28 days prior to Study Day 0
* Patients who meet the following laboratory parameter:

  * Lymphocyte count >= 1000 cells/mm³
  * Hemoglobin >= 9.0 g/dl (men and women)
  * Platelet count >= 75000 cells/mm3
  * Alkaline Phosphatase <= 3.0 times the upper limit of normal
  * Serum Glutamic-Oxaloacetic Transaminase (SGOT) and Serum Glutamic-Pyruvic Transaminase (SGPT) <= 3.0 times the upper limit of normal
  * Total bilirubin <= 1.5 times the upper limit of normal
  * Creatinine <= 2mg/dL
* Female patients of reproductive potential must be willing to use a reliable method of double-barrier contraception (such as diaphragm with spermicidal cream or jelly, or condoms with spermicidal foam)
* Patients who are informed of and willing and able to comply with the investigational nature of the study and had signed a written consent in accordance with institutional and federal guidelines
* Patients who have been on stable antiretroviral therapy (no changes in medication or dose) for at least thirty days prior to study entry and who will continue on background during study participation

Exclusion Criteria:

* Female patients who are pregnant or breast-feeding
* Patients requiring systemic treatment with corticosteroids or drugs known to be hepatic enzyme inducers or inhibitors within 14 days of stud entry (Study Day 0). Such substances in these categories include: macrolide antibiotics (erythromycin, clarithromycin), azole antifungals (ketoconazole, fluconazole, itraconazole) rifampin, rifabutin, and phenytoin
* Patients receiving any investigational drug within 30 days of the first dose of study medication and any antineoplastic agent or radiotherapy other than local skin radiotherapy treatment within 12 weeks before starting study medication
* Patients with malabsorption, severe chronic diarrhea or patients unable to maintain adequate oral intake
* Patients with a history of intravenous drug abuse, alcohol or substance abuse considered by the Investigator and Boehringer Ingelheim Pharmaceutical Incorporated (BIPI) Medical Monitor to be a significant impairment to health and compliance
* Patients undergoing treatment for an active infection
* Patients with hepatic insufficiency due to cirrhosis
* Patients with renal insufficiency
* Patients who are heavy smokers (e.g. > 20 cigarettes per day)
* Patients currently taking Norvir® (Ritonavir) or Rescriptor® (Delavirdine)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 1998-04; Primary Completion 1999-04 (Actual)

PRIMARY OUTCOMES:
AUC (Area under the plasma concentration time curve) of ethinyl estradiol/norethindrone (EE/NET) | 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 15, 24, and 34 hours post dose on day 0 and day 30
Cmax (maximum observed concentration) of EE/NET | 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 15, 24, and 34 hours post dose on day 0 and day 30
Tmax (Time of maximum concentration) of EE/NET | 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 15, 24, and 34 hours post dose on day 0 and day 30
AUCss (Area under the concentration time curve at steady state) of nevirapine | 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 15, 24, and 34 hours post dose on day 30
Cmax (maximum observed concentration) of nevirapine | 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 15, 24, and 34 hours post dose on day 30
Cmin (minimum observed concentration) of nevirapine | 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 15, 24, and 34 hours post dose on day 30
Cl/F (Oral clearance) of nevirapine | 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 15, 24, and 34 hours post dose on day 30

SECONDARY OUTCOMES:
Number of patients with adverse events | up to 59 days